CLINICAL TRIAL: NCT05223465
Title: Faculty and Students' Attitude Toward E-learning at the Start of the COVID-19 Pandemic: A Cross-sectional Study
Brief Title: Faculty and Students' Attitude Toward E-learning
Status: Completed | Type: Observational
Sponsor: Hawler Medical University (Other)
Responsible Party: Principal Investigator, Nazdar Ezzaddin Alkhateeb, Assistant Professor, Hawler Medical University
Other Study IDs: 412312022
Record Dates: First submitted 2022-01-19; First posted 2022-02-04 (Actual); Last update posted 2022-02-04 (Actual); Status verified 2022-01

CONDITIONS: E Learning; Medical Education
Keywords: Medical Education; E-learning; COVID-19; Students' attitude; Facultys' attitude
MeSH Terms: conditions — COVID-19 | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Survey — Google form distributed for students and faculties

SUMMARY:
E-learning in medical education is a relatively new idea that is rapidly growing. This study aimed to assess the students and faculty staff attitude for e-learning at the emergence of COVID-19.

A prospective cross-sectional online survey based on Google form was conducted at a medical university in Iraq between March and April 2020

DETAILED DESCRIPTION:
E learning provides education at a generally lower cost and engages learners at a time and location that is most appropriate for them. Recent calls for reform in medical education and training have emphasized the use of information technology-empowered learning. This was enhanced more in the COVID-19 era . Some international organizations, such as the World Health Organization (WHO), have acknowledged e-learning as a helpful tool for healthcare education, particularly in developing countries. Nevertheless, the use of e-learning by the faculty members and students stayed minimum for uploading lecture notes, course books, feedbacks, and providing marks until the COVID-19 pandemic raised that need. This study aimed to evaluate faculty and students' knowledge and attitudes toward e-learning at the emergence of COVID-19 and identify the potential requirements for implementing e-learning.

An online survey was distributed to a sample of 190 faculty and 1706 students of a medical university in Iraq. Knowledge and attitudes towards e-learning were studied

ELIGIBILITY:
Inclusion Criteria:

* undergraduate students faculty staff working in Hawler Medical University

Exclusion Criteria:

* Faculty staff who are on leave for study or health purpose

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The population is composed of students studying in colleges of Haler Medical University (Medicine, Dentistry, Pharmacy, nursing and health science) in addition to faculty staff working in the above-mentioned colleges
Sampling Method: Non-Probability Sample
Enrollment: 1896 (Actual)
Dates: Start 2020-03-01 (Actual); Primary Completion 2020-04-30 (Actual); Study Completion 2021-06-30 (Actual)

PRIMARY OUTCOMES:
Knowledge | At the beginning of the study
  Students and faculties response collected on their knowledge about e-learning
Attitude | At the beginning of the study
  Students and faculties response collected on their Attitude about e-learning

SECONDARY OUTCOMES:
Opinion | At the beginning of the study
  faculties and students opinion on alternative ways for assessment

CONTACTS AND LOCATIONS:
Overall Officials: Nazdar E Alkhateeb, PhD, Principal Investigator — Hawler Medical University
Locations (1):
- Nazdar Ezzaddin Alkhateeb, Erbil, Kurdistan Region, Iraq

IPD SHARING:
Plan to Share IPD: Undecided